CLINICAL TRIAL: NCT00462579
Title: Risk Factors for Carbapenem-resistant Acinetobacter Baumannii
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: PRO07040057
Record Dates: First submitted 2007-04-17; First posted 2007-04-19 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Acinetobacter Infections
Keywords: carbapenem-resistant acinetobacter baumannii; positive culture; positive culture for carbapenem-resistant acinetobacter
MeSH Terms: conditions — Acinetobacter Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
It has been demonstrated that panresistant strains of Acinetobacter species may be selected by antibiotic use [4], may be transmitted from person to person [5], and may be passed via environmental contamination [6]. Surveillance for panresistant Acinetobacter species should be a priority, given the lack of antibiotic options for the treatment of these infections. There are currently no data on the antibiotic susceptibility of Acinetobacter species or on the rates of panresistant organisms. The elucidation of potential risk factors for resistant strains of Acinetobacter is therefore an important task, and the use of alternative antibiotics should be considered in ICUs where these strains are endemic.

DETAILED DESCRIPTION:
The elucidation of potential risk factors for resistant strains of Acinetobacter is therefore an important task, and the use of alternative antibiotics should be considered in ICUs where these strains are endemic.he following information will be collected: age, sex, occupation, hospital location at the time of positive culture (ER, medical ward, ICU etc), date of positive culture, prior hospitalization, receipt of outpatient dialysis, home care or other regular medical care (eg, outpatient chemotherapy), presence of invasive devices, receipt of antibiotics, including their type and whether they were adequate for the resistance profile of the organism, prior positive microbiologic cultures, time and location of positive cultures, underlying diseases and severity of illness, presence of urinary or intravascular devices, recent immunomodulative therapies or radiation therapy, physical exam findings, laboratory and radiographical data, antimicrobial usage within 30 days of onset of the infection, microbiological data and resistance patterns, choice of antibiotics once organism identified, bacteriological outcomes, laboratory results, demographic information, medications, clinical outcome,gender, height, weight, ethnicity, and past medical history. We will collect information retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Positive cultures of carbapenem-resistant acinetobacter baumannii

Exclusion Criteria:

* Not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: carbapenem-resistant acinetobacter baumannii positive cultures
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-04 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
dead or alive | end of study
  health status

CONTACTS AND LOCATIONS:
Overall Officials: David L Paterson, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States